CLINICAL TRIAL: NCT03644030
Title: Comparative Assessment of Phase Angle, Lean Body Mass Index and Tissue Edema to Assess the Nutritional Status and Immediate Outcome of Cardiac Surgery Patients:an Open, Prospective Study of Observation / Recording
Brief Title: Phase Angle, Lean Body Mass Index and Tissue Edema and Immediate Outcome of Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, katerina kotzampassi, Surgeon Director of NSI, Aristotle University Of Thessaloniki
Other Study IDs: CardioMass
Record Dates: First submitted 2018-08-11; First posted 2018-08-23 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2018-09

CONDITIONS: Sarcopenia; Post-operative Infections; Sepsis
Keywords: FFM index; tissue edema index [extracellular / total water - ECW / TBW]; phase angle
MeSH Terms: conditions — Sarcopenia; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In general, malnutrition in surgical patients is associated with a higher risk of postoperative infections, decreased immune response, more cardiac complications, prolonged mechanical ventilation , and a higher rate of reimportation due to several other complications than lead to an increase in morbidity and mortality, a prolongation of the total hospitalization time in the ICU[intensive care unit ] and the chamber, and a delay in the healing of the surgical trauma .

The presence of a low percentage of lean mass, as calculated by the technique of bioelectric conductivity, practically means a small percentage of muscle tissue. However, muscle tissue is an important, if not the only source of amino acids for both protein synthesis and gluconeogenesis in stress conditions, such as surgery and the first postoperative days. Thus, post-operative patients in general, and cardio-operated patients, in particular, having a low lean mass have minimal reserves to the stress requirements, resulting in an increased risk of complications.

In the last few years, the most reliable indicator of malnutrition- in addition to the lean mass index - began to be considered the phase angle, which is also calculated when measuring the bioreduction of electrical conductivity, although there is a very recent challenge . The phase angle expresses the relationship between the electrical reactance, i.e. the state of the cell membrane, to resist the permeability and the resistance, i.e. the restriction to the flow of the electrical current through the body, mainly related to the water of the tissues . Like the FFM[fat-free mass]- index, the phase angle uses the total water of the tissues, and thus also reflects the cell mass. In addition, however, it also measures the resistance of cell membranes, so it also evaluates their quality and is therefore considered to be a reliable indicator of poor nutritional status , although some also maintain demur due to the possible poor distribution of extracellular fluid in cardiological patients.

From all of the above, it appears that there are some gaps in the evaluation of the patients who are going to undergo cardiac surgery regarding their nutritional status, both because the classic nutrition control indicators are not fully documented as being reliable for these patients, and there are no studies to monitor and compare body composition directly to any other index postoperatively.

DETAILED DESCRIPTION:
The study protocol-mandated baseline data will include demographics, comorbidities, EuroSCORE[European System for Cardiac Operative Risk Evaluation] II, C-reactive protein, left ventricular ejection fraction (by transthoracic echocardiography) and peak expiratory flow rate (assessed by spirometry). Physical performance status will be assessed by APACHE [Acute Physiology And Chronic Health Evaluation] II score. Furthermore, SOFA [Sequential [Sepsis-related] Organ Failure Assessment] score will be assessed preoperatively and up to 7th postoperative day.

Preoperatively and on the 7th postoperative day, the following parameters will be calculated or measured and then recorded:

* Anthropometric data including body height, weight and waist circumference measurement, estimation of waist/circumference ratio and calculation of body mass index [BMI].
* Nutritional status will be assessed by MUST[Malnutrition Universal Screening Tool] score
* Body composition analysis using bioelectrical impedance analysis [BIA], will be performed for the calculation of FFM [fat-free mass] and fat mass [FM] indicators, intracellular, extracellular and total water [ICW, ECW, TBW] and phase angle parameter [PhA]. Additionally, muscular power will be assessed by handgrip strength [HGS], the upper third triangle perimeter and skin fold thickness will be measured.
* Daily calorie and protein needs of each patient will be calculated

During hospitalization, the following parameters will be recorded:

* Type of diet [parenteral, intestinal, oral]
* Post-operative infections involving respiratory system, medieval space, sternum trauma, lower limb trauma (if present) and endocarditis.
* The occurrence of organ dysfunction or sepsis. Sepsis is defined as a life-threatening organ dysfunction caused by a dysregulated host response to infection. For clinical operationalization, organ dysfunction will be represented by an increase in the Sequential [Sepsis-related] Organ Failure Assessment (SOFA) score of 2 points or more, which will be associated with an in-hospital mortality greater than 10%.
* Thromboembolic events such as stroke, peripheral venous thrombosis and pulmonary embolism.
* Acute renal failure.
* Re-operation for bleeding.
* Need for inotropic or vasoactive support.
* Hospitalization data (intubation> 24 hours, duration of mechanical ventilation and ICU stay, duration of hospital stay, in-hospital mortality

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* planned introduction for cardiac operation with CPB[cardiopulmonary bypass]
* coronary artery bypass surgery
* heart valve surgery [heart valve surgery]

Exclusion Criteria:

* non-consent of the patient
* urgent admissions - operations
* pacemaker exist
* congenital heart disease
* recent [<3-month] open-heart surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo cardiac surgery for coronary revascularization or valvular heart disease
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Phase angle in patients undergoing cardiac surgery as indicator of their nutrition status. | 7 days post operation
  Phase angle [PhA(°) = (reactance/electrical resistance) × (180°/Π)] will be measured in degrees using bioelectrical impedance analysis and check whether it can be considered as a reliable indicator of the nutrition status of cardiac surgery patients undergoing cardiac surgery during the preoperative and postoperative periods. PhA will be calculated by using the sum of impedance and reactance of the right arm, trunk, and right leg and based on the following equation, PhA(°) = (Reactance/Resistance) × (180°/Π). Π is the mathematical value of 3.1415 and This conversion is performed to convert the final value from radians into degrees.The normal range of phase angle is 5.84 ± 0.75.The primary change is the reduction of the mean phase angle postoperative by 1.0 unit (standard deviation ± 2.0) and this leads to increased morbidity, mortality.

SECONDARY OUTCOMES:
FFM[fat-free mass] index(kilograms/(meter x meter)- kg/m-2) in patients undergoing cardiac surgery as indicator of their nutrition status | 7 days post operation
  measure of FFM [fat-free mass] index( kgm-2) using bioelectrical impedance analysis and check if it can be a reliable indicator of the nutrition status of patients undergoing cardiac surgery during the preoperative and post-operative periods and how this leads to increased morbidity, mortality.
Tissue edema index [extracellular(Litre) / total water(Litre) - ECW / TBW] in patients undergoing cardiac surgery as indicator of their nutrition status. | 7 days post operation
  measure of the tissue edema index [extracellular(Litre) / total water(Litre) - ECW / TBW] using bioelectrical impedance analysis and check if it can be a reliable indicator of the nutrition status of patients undergoing cardiac surgery during the preoperative and post-operative periods and if this associated with postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Kotzampassi, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Visser M, van Venrooij LM, Vulperhorst L, de Vos R, Wisselink W, van Leeuwen PA, de Mol BA. Sarcopenic obesity is associated with adverse clinical outcome after cardiac surgery. Nutr Metab Cardiovasc Dis. 2013 Jun;23(6):511-8. doi: 10.1016/j.numecd.2011.12.001. Epub 2012 Mar 6. PMID 22397879
- [Background] Lomivorotov VV, Efremov SM, Boboshko VA, Nikolaev DA, Vedernikov PE, Deryagin MN, Lomivorotov VN, Karaskov AM. Prognostic value of nutritional screening tools for patients scheduled for cardiac surgery. Interact Cardiovasc Thorac Surg. 2013 May;16(5):612-8. doi: 10.1093/icvts/ivs549. Epub 2013 Jan 29. PMID 23360716
- [Background] Gomez-Perez SL, Haus JM, Sheean P, Patel B, Mar W, Chaudhry V, McKeever L, Braunschweig C. Measuring Abdominal Circumference and Skeletal Muscle From a Single Cross-Sectional Computed Tomography Image: A Step-by-Step Guide for Clinicians Using National Institutes of Health ImageJ. JPEN J Parenter Enteral Nutr. 2016 Mar;40(3):308-18. doi: 10.1177/0148607115604149. Epub 2015 Sep 21. PMID 26392166
- [Background] Tsaousi G, Panidis S, Stavrou G, Tsouskas J, Panagiotou D, Kotzampassi K. Prognostic indices of poor nutritional status and their impact on prolonged hospital stay in a Greek university hospital. Biomed Res Int. 2014;2014:924270. doi: 10.1155/2014/924270. Epub 2014 Mar 23. PMID 24779021
- [Background] van Venrooij LM, de Vos R, Borgmeijer-Hoelen MM, Haaring C, de Mol BA. Preoperative unintended weight loss and low body mass index in relation to complications and length of stay after cardiac surgery. Am J Clin Nutr. 2008 Jun;87(6):1656-61. doi: 10.1093/ajcn/87.6.1656. PMID 18541553
- [Background] van Venrooij LM, de Vos R, Zijlstra E, Borgmeijer-Hoelen MM, van Leeuwen PA, de Mol BA. The impact of low preoperative fat-free body mass on infections and length of stay after cardiac surgery: a prospective cohort study. J Thorac Cardiovasc Surg. 2011 Nov;142(5):1263-9. doi: 10.1016/j.jtcvs.2011.07.033. Epub 2011 Aug 19. PMID 21855896
- [Background] Visser M, van Venrooij LM, Wanders DC, de Vos R, Wisselink W, van Leeuwen PA, de Mol BA. The bioelectrical impedance phase angle as an indicator of undernutrition and adverse clinical outcome in cardiac surgical patients. Clin Nutr. 2012 Dec;31(6):981-6. doi: 10.1016/j.clnu.2012.05.002. Epub 2012 May 27. PMID 22640476
- [Background] Tsaousi G, Kokkota S, Papakostas P, Stavrou G, Doumaki E, Kotzampassi K. Body composition analysis for discrimination of prolonged hospital stay in colorectal cancer surgery patients. Eur J Cancer Care (Engl). 2017 Nov;26(6). doi: 10.1111/ecc.12491. Epub 2016 Mar 16. PMID 26990464
- [Background] Engelman DT, Adams DH, Byrne JG, Aranki SF, Collins JJ Jr, Couper GS, Allred EN, Cohn LH, Rizzo RJ. Impact of body mass index and albumin on morbidity and mortality after cardiac surgery. J Thorac Cardiovasc Surg. 1999 Nov;118(5):866-73. doi: 10.1016/s0022-5223(99)70056-5. PMID 10534692
- [Background] van Straten AH, Bramer S, Soliman Hamad MA, van Zundert AA, Martens EJ, Schonberger JP, de Wolf AM. Effect of body mass index on early and late mortality after coronary artery bypass grafting. Ann Thorac Surg. 2010 Jan;89(1):30-7. doi: 10.1016/j.athoracsur.2009.09.050. PMID 20103201
- [Background] Wagner BD, Grunwald GK, Rumsfeld JS, Hill JO, Ho PM, Wyatt HR, Shroyer AL. Relationship of body mass index with outcomes after coronary artery bypass graft surgery. Ann Thorac Surg. 2007 Jul;84(1):10-6. doi: 10.1016/j.athoracsur.2007.03.017. PMID 17588373
- [Background] Soeters PB, Schols AM. Advances in understanding and assessing malnutrition. Curr Opin Clin Nutr Metab Care. 2009 Sep;12(5):487-94. doi: 10.1097/MCO.0b013e32832da243. PMID 19512916